CLINICAL TRIAL: NCT05869071
Title: Agreement Between Accelerometric and Acoustic Signals Utilizing Algorithm and Body Plethysmograph in Detecting Nasal and Oral Specific Airway Resistance
Brief Title: Assessment of Oral and Nasal Breathing With Sensors Analyzing Algorithm
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Olli-Pekka Alho, MD, Professor, Oulu University Hospital
Other Study IDs: 126/2021
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Nasal Polyps; Asthma; COPD; Allergic Rhinitis
MeSH Terms: conditions — Nasal Polyps; Asthma; Pulmonary Disease, Chronic Obstructive; Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy volunteers: Participants with no chronic disease and no acute symptoms
  Interventions: Device: Sensor analyzing software (own development); Device: Body plethysmograph
- Patients with Allergic rhinitis or Nasal Polyps: Participants with allergic rhinitis or nasal polyps
  Interventions: Device: Sensor analyzing software (own development); Device: Body plethysmograph
- Patients with asthma: Participants with asthma
  Interventions: Device: Sensor analyzing software (own development); Device: Body plethysmograph
- Patients with COPD: Participants with Chronic Obstructive Pulmonary Disease
  Interventions: Device: Sensor analyzing software (own development); Device: Body plethysmograph

INTERVENTIONS:
Device: Sensor analyzing software (own development) — A software the research group developed. Analyzes acoustic and accelerator signals to measure airway obstruction.
Device: Body plethysmograph — Body plethysmograph measures specific airway resistance
  Other Names: Ganshorn PowerCube body+ plethysmograph

SUMMARY:
The goal of this observational study is to learn about the agreement between sensors analyzing algorithm and body plethysmography in measuring oral and nasal breathing in healthy adults, and in patients with chronic rhinosinusitis, asthma and chronic obstructive pulmonary disease. The main question it aims to answer is: • Is the algorithm-based method accurate enough in analyzing respiratory obstruction as compared to body plethysmography (reference method)? Participants will perform a short breathing protocol (oral and nasal breathing with different masks) during which time their breathing is monitored with both methods.

DETAILED DESCRIPTION:
The data collected in the Patient Registry include: Parameters on general health, like previous illnesses, medications, height, weight, answers to symptoms queries and queries on quality of life (Asthma test, COPD test, Sinonasal Outcome Test 22) as well as results from the examined medical devices (body plethysmography, spirometry, sensors analyzing algorithm).

ELIGIBILITY:
Inclusion Criteria:

* 5 healthy and asymptomatic volunteers with regard to lungs and nose
* 5 patients with allergic rhinitis or nasal polyps (diagnosis of allergic rhinitis confirmed by a PRICK test or specific Ig E antibody tests and Nasal polyposis diagnosed by an ENT specialist, with endoscopy)
* 5 patients with asthma (diagnosis of asthma based on peak expiratory flow (PEF) monitoring, spirometry, or other appropriate objective measurement methods performed by a pulmonologist
* 5 patients with Chronic Obstructive Pumonary Disease (diagnosis of COPD based on spirometry (post-bronchodilator Forced Expiratory Volume/ Forced Vital Capacity (FEV1/FVC) ratio below 0.70)

Exclusion Criteria:

* Pregnancy.
* History of surgical procedures in the chest, larynx, throat (excluding tonsillectomy), or nasal area.
* Recent illnesses or surgeries that pose a risk to the patient or prevent proper measurement (common contraindications for spirometry):
* Recent (<1 month) myocardial infarction.
* Severe coronary artery disease with easily triggered symptoms.
* Cerebral artery aneurysm.
* Recent brain (<4 weeks) or eye (<1 week) surgery.
* Severe cardiac arrhythmias.
* Pulmonary tuberculosis.
* Pneumothorax
* Immediate postoperative period of lung surgery (<1 day).
* Dementia or confusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The healthy volunteers are selected from the personnel or students of Oulu University Hospital and University of Oulu. The patients with allergic rhinitis and nasal polyps, asthma and Chronic Obstructive Pulmonary Disease are selected from the Oulu University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Bias for oral breathing (estimate and 95% confidence intervals) | 5 minutes
  Bias between specific airway resistances given by analyzing software and plethysmograph
Bias for nasal breathing (estimate and 95% confidence intervals) | 5 minutes
  Bias between specific airway resistance given by analyzing software and plethysmograph
Limits of agreement for oral breathing | 5 minutes
  Limits of agreement between specific airway resistance given by analyzing software and plethysmograph
Limits of agreement for nasal breathing | 5 minutes
  Limits of agreement between specific airway resistance given by analyzing software and plethysmograph

SECONDARY OUTCOMES:
Mean error for oral breathing (estimate and 95% confidence intervals) | 5 minutes
  Mean error between specific airway resistance given by analyzing software and plethysmograph
Mean error for nasal breathing (estimate and 95% confidence intervals) | 5 minutes
  Mean error between specific airway resistance given by analyzing software and plethysmograph
Correlation between analyzing software and subjective sensation of oral breathing obstruction | 5 minutes
  Correlation between specific airway resistance and graded (6 steps) subjective sensation
Correlation between analyzing software and subjective sensation of nasal breathing obstruction | 5 minutes
  Correlation between specific airway resistance and graded (6 steps) subjective sensation
Correlation between plethysmograph and subjective sensation of oral breathing obstruction | 5 minutes
  Correlation between specific airway resistance and graded (6 steps) subjective sensation
Correlation between plethysmograph and subjective sensation of nasal breathing obstruction | 5 minutes
  Correlation between specific airway resistance and graded (6 steps) subjective sensation
Reliability of analyzing software measurement | 5 minutes
  Measurer's opinion of the reliability of the measurement (4 steps)
Reliability of plethysmograph | 5 minutes
  Measurer's opinion of the reliability of the measurement (4 steps)
Convenience of analyzing software method | 5 minutes
  Metrizable's opinion of the convenience (6 steps)
Convenience of plethysmography | 5 minutes
  Metrizable's opinion of the convenience (6 steps)
Harms of analyzing software method | 5 minutes
  Frequency of harmful events related to measurement
Harms of plethysmography | 5 minutes
  Frequency of harmful events related to measurement

CONTACTS AND LOCATIONS:
Overall Officials: Olli-Pekka Alho, Prof, Principal Investigator — University of Oulu, Finland
Locations (1):
- Oulu University Hospital, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No